CLINICAL TRIAL: NCT01349738
Title: Asymptomatic Bacteriuria & Risk of Urinary Tract Infection in Renal Transplants
Acronym: ASB
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rice, James C., M.D. (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Dr. James C. Rice, Scripps
Other Study IDs: ASB in Transplants
Record Dates: First submitted 2011-05-04; First posted 2011-05-09 (Estimated); Last update posted 2011-09-01 (Estimated); Status verified 2011-08

CONDITIONS: Bacteriuria; Urinary Tract Infections; Asymptomatic Infections; Transplantation Infection
MeSH Terms: conditions — Bacteriuria; Urinary Tract Infections; Asymptomatic Infections | interventions — Anti-Bacterial Agents; Trimethoprim, Sulfamethoxazole Drug Combination; Levofloxacin; Ampicillin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The investgators have a repository of bacteria specimens from transplant patients with UTI and plan to save bacteria from this study. The investigators will also plan to save discarded aliquots of supernatent of urine and discarded aliquots of blood, all samples from centrifuged specimens devoid of human cells.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Positive Group: Positive for ASB
  Interventions: Drug: Antibiotic
- Negative Group: Negative for ASB

INTERVENTIONS:
Drug: Antibiotic — Antibiotic (drug) sensitive to most recent culture for these subjects testing ASB positive and also experience Signs and symptoms of a UTI
  Other Names: Trimethoprim sulfamethoxazole (Bactrim); Levofloxacin (Levaquin); Ampicillin; SUSCEPTIBILITY; Organism >100,000 col/ml Escherichia coli (presumptive); Susceptibility type MIC (BY VITEK 2); Ampicillin >=32 Resistant; Ampicillin/Sulbactam 16 Intermediate; Cefazolin <=4 Suscep.; Ciprofloxacin <=0.25 Suscep.; Gentamicin <=1 Suscep.; Levofloxacin <=0.12 Suscep.; Nitrofurantoin <=16 Suscep.; Tobramycin <=1 Suscep.; Trimeth-Sulfa >=16/304 Resistant
  Groups: Positive Group

SUMMARY:
The goal of this research program is to understand the natural history of asymptomatic bacteriuria in the renal transplant patients, to determine if screening for asymptomatic bacteriuria and identification of key host characteristics and virulence factors present on uropathogenic bacteria identifies a sub-population of patients with asymptomatic bacteriuria that are at risk to develop symptomatic urinary tract infection. Ultimately, the knowledge obtained from this study will prevent inappropriate antibiotic use and may identify whether certain bacterial isolates predispose to renal allograft injury. We will test the hypothesis that (i) asymptomatic bacteriuria is common in the renal allograft recipient and (ii) that symptomatic urinary tract infection and renal allograft dysfunction do not occur unless key host susceptibility factors and uropathogenic bacterial virulence factors are present.

DETAILED DESCRIPTION:
Blood samples and urine cultures will be obtained from asymptomatic renal transplant clinic patients. If the urine culture is positive (> or = 105 cfu/ml), we will determine the host and bacterial virulence factors associated with asymptomatic bacteriuria (ASB) and compare these results to transplant patients that develop a symptomatic UTI. The patient's clinical information, laboratory data and the bacterial isolate responsible for the UTI will be collected at the time of their clinic visit and subsequently analyzed.

After the first visit (Day 0 after signing consent) blood and urine will be collected, subjects will be put into either ASB Positive or ASB Negative groups based upon the results of their urine culture. From that point, those who test into the ASB Negative group will have an additional urine culture, either by returning to the clinic or by sending a urine culture mailer kit, and if cultures remain negative, they will be discharged from the study after reviewing medications, adverse events and completing a urinary tract infection risk questionnaire.

For those who test into the ASB Positive group, those subjects will be monitored by the subject returning to the clinic on Day 10-14, at 1 month, 2 month, 3 month and 6 months for blood and urine collection, review of medications and adverse events, and completing a urinary tract infection risk questionnaire. Should the subject have symptoms of a UTI, the subject will be treated with the appropriate antibiotic for which the bacterial isolated from their urine culture is sensitive. Patients will return to the clinic 10-14 days later for a repeat urine culture, complete a urinary tract infection risk questionnaire, and have a repeat urine culture to confirm they are urinary tract infection free. At this point, the subject will be discharged from the study after reviewing medications and adverse events.

It is predicted that 75% of patients will test into the ASB Negative Group and do not require antibiotic therapy. We predict that 25% of patients will test into the ASB Positive Group, but that less than 5% of these patients will ultimately develop a symptomatic UTI and require antibiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* must be 18 years old or older,
* had a kidney transplant,
* be at least 30 days post operation.

Exclusion Criteria:

* Pregnant women, those planning to become pregnant or nursing mothers;
* Renal transplant patients less than 30 days post transplant; Use of an indwelling Foley catheter;
* Patients without a renal transplant;
* Patients having concurrent surgical/wound infection and presumed hematogenous dissemination for the urinary tract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney Transplant Patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-05; Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Asymptomatic Bacteriuria and Risk of Developing Symptomatic Urinary Tract Infections or Renal Allograft Injury in Renal Transplant Patients | 2 years
  Determine the prevalence and natural history of asymptomatic bacteriuria (ASB) and the host factors associated with the development of symptomatic UTI in renal allograft recipients. We will enroll renal transplant recipients, perform urine cultures and follow all patients with ASB to determine the prevalence of ASB and the host characteristics associated with ASB and the development of symptomatic UTI.

SECONDARY OUTCOMES:
Host Characteristics of Renal Transplant Patients with Asymptomatic Bacteriuria at Risk to Develop Symptomatic Urinary Tract Infection | 2 years
  We will measure blood and urine immunoglobulin and cytokine levels in patients with ASB and symptomatic UTI to determine if these host's immune parameters predict the outcome of ASB, including the development of symptomatic UTI.
Determine the characteristics of uropathogenic bacteria that cause acute allograft injury in renal transplant patients. | 2 years
  We will determine the expression of key uropathogenic virulence factors, including P fimbriae, Dr adhesins, and mono-mannose-binding type 1 fimbriae, on E. coli isolated from RTPs with ASB to determine if strains that express such virulence factors are more likely to cause symptomatic UTI and AAI, compared to E. coli that do not express these virulence factors.

CONTACTS AND LOCATIONS:
Overall Officials: James C. Rice, MD, Principal Investigator — Scripps
Locations (1):
- Scripps Green Hospital, La Jolla, California, United States